CLINICAL TRIAL: NCT04722133
Title: A Phase II Trial of Trastuzumab-pkrb Combined With Modified FOLFOX-6 in Biliary Tract Cancer Patients Progressed on First Line Therapy
Brief Title: Trastuzumab-pkrb Combined With Modified FOLFOX-6 in Biliary Tract Cancer Patients Progressed on First Line Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-0648
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: HER2 Positive Advanced/Metastatic/Nonresectable Biliary Tract Cancer
Keywords: biliary tract cancer; HER2; herzuma; trastuzumab
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HERZUMA+mFOLFOX (Experimental)
  Interventions: Drug: HERZUMA+mFOLFOX

INTERVENTIONS:
Drug: HERZUMA+mFOLFOX — Herzuma (Trastuzumab-pkrb) 4mg/kg after 6mg/kg loading D1 5FU 400mg/m2 bolus+2400mg/m2 infusion for 46 hrs D1 Leucovorin 200mg/m2 D1 Oxaliplatin 85mg/m2 D1 every 2 weeks

SUMMARY:
Trastuzumab is approved for the treatment of HER2-positive breast cancer and gastric cancer. The recent study showed that HER2 overexpression or amplification is noted about 5-15% of total biliary tract cancer patients and have shown efficacy in small basket trials. The aim of this study is to evaluate the efficacy and safety of trastuzumab in the combination of mFOLFOX for gemcitabine+cisplatin refractory biliary tract cancer patients.

DETAILED DESCRIPTION:
This phase II study is designed to see whether trastuzumab-pkrb+FOLFOX is active as 2nd or 3rd line treatment for HER2-positive biliary tract cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented recurred/metastatic/unresectable biliary tract cancer, including gallbladder cancer, intrahepatic, extrahepatic cholangiocarcinoma, or ampulla of vater cancer.
2. Histologically confirmed HER2 positive biliary tract cancer. HER2-positive tumor was defined as either IHC 3+ or IHC 2+ in combination with ISH +, or ERBB2 amplification (≥6 copies) by tumor tissue NGS.
3. Recurred/metastatic/unresectable biliary tract cancer patient whose disease progression was confirmed by imaging modality after gemcitabine+cisplatin containing 1st line palliative chemotherapy regimen. Previous lines should be one or two (immunotherapy monotherapy not counted).
4. be willing and able to provide written informed consent/assent for the trial
5. be at least 19 years of age on day of signing informed consent
6. have measurable disease based on RECIST (Response Evaluation Criteria In Solid Tumors) version 1.1
7. have a performance status of 0 or 1 on the ECOG (Eastern Cooperative Oncology Group) Performance Scale
8. demonstrate adequate organ function
9. No severe valvular or arrhythmic cardiac disease with LVEF ≥ 50%
10. female subject of childbearing potential should have a negative urine or serum pregnancy or be willing to use birth control

Exclusion Criteria:

1. Previous treatment history of oxaliplatin containing chemotherapy, anti-HER2 targeting treatment (trastuzumab, neratinib, lapatinib, and etc)
2. has had a prior anti-cancer chemotherapy, targeted small molecule therapy, or radiotherapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered.
3. has a known additional malignancy that is progressing or requires active treatment within 3 years, except basal cell carcinoma of the skin, squamous cell carcinoma of the skin and thyroid cancer that has undergone potentially curative therapy or in situ cervical cancer
4. has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
5. has known history or evidence of any disease, treatment, or laboratory results that would inhibit the patient's participation to the study.
6. Has clinically significant cardiac disease, including congestive heart failure ≥ NYHA grade 2, uncontrolled hypertension, QTcF > 470 msec or QT prolong syndrome, recent myocardiac infarction or unstable angina history
7. has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
8. is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
9. has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
10. has known active Hepatitis B (HBsAg reactive and HBV DNA 100 ≥copies/ml) or Hepatitis C (anti-HCV reactive and HCV RNA [qualitative] is detected)
11. has received a live vaccine within 30 days of planned start of study therapy.
12. has an active infection requiring systemic therapy
13. has history of severe adverse event or allergic reaction to 5-FU, leucovorin, oxaliplatin or trastuzumab
14. need O2 supply or show dyspnea on rest due to advanced malignancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  rate of patients with complete remission (CR) or partial remission (PR) based on RESIST1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 2 years
  PFS is defined as time interval from cycle 1 day 1 to tumor progression/death/last follow-up
Disease control rate (DCR) | up to 2 years
  DCR is rate of patients with CR, PR, or SD per RECIST 1.1.
Overall survival (OS) | up to 2 years
  OS is defined as time interval from cycle 1 day 1 to tumor death/last follow-up.
Incidence of treatment related adverse events (TRAE) | up to 2 years
  Incidence of treatment related adverse events (TRAE) will be assessed using NCI CTCAE v5.0 and tabulated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Choong-kun Lee, Principal Investigator — Severance Hospital
Locations (1):
- Division of Medical Oncology, Yonsei Cancer Center, Yonsei Univ. College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee CK, Chon HJ, Cheon J, Lee MA, Im HS, Jang JS, Kim MH, Park S, Kang B, Hong M, Kim JW, Park HS, Kang MJ, Park YN, Choi HJ. Trastuzumab plus FOLFOX for HER2-positive biliary tract cancer refractory to gemcitabine and cisplatin: a multi-institutional phase 2 trial of the Korean Cancer Study Group (KCSG-HB19-14). Lancet Gastroenterol Hepatol. 2023 Jan;8(1):56-65. doi: 10.1016/S2468-1253(22)00335-1. Epub 2022 Oct 31. PMID 36328033